CLINICAL TRIAL: NCT02033486
Title: Digital Breast Tomosynthesis Guided Tomographic Optical Breast Imaging (TOBI)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mansi A Saksena, Assistant Professor at Massachusetts General Hospital, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013P000488; 5R01CA142575 (NIH); R01CA187595 (NIH)
Record Dates: First submitted 2014-01-09; First posted 2014-01-10 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer
Keywords: diffuse optical tomography; digital breast tomosynthesis; breast cancer; solid benign lesions; cysts; malignant lesions
MeSH Terms: conditions — Breast Neoplasms; Cysts | interventions — Mammography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TOBI + DBT (Experimental): TOBI + DBT of women presenting for breast imaging.
  Interventions: Device: TOBI + DBT

INTERVENTIONS:
Device: TOBI + DBT
  Other Names: Diffuse Optical Tomography + digital breast tomosynthesis

SUMMARY:
Screening for breast cancer improves early detection of aggressive cancers and has been shown to reduce breast cancer related mortality. Currently, mammography is the most effective way of detecting early stage, non palpable breast cancers. However, mammography only reveals the breast structure, and cannot say much about the breast physiological state. We propose Tomographic Optical Breast Imaging (TOBI) as an inexpensive, patient friendly technique that is non-invasive and does not use non-ionizing radiation. TOBI uses near infrared light and by measuring how such light passes through the breast, images of blood volume and hemoglobin oxygenation can be obtained. In this study, TOBI is combined with digital breast tomosynthesis (DBT, a form of 3D mammography) and our hypothesis is that the TOBI-DBT combined images can be used to diagnose breast cancer with significantly improved sensitivity and specificity compared to DBT alone.

ELIGIBILITY:
Inclusion Criteria:

* Any adult female volunteers of any race or ethnic background, between the ages of 30 to 80, either

  * scheduled for a clinically indicated diagnostic mammogram or percutaneous biopsy.
  * presenting for breast cancer treatment

Exclusion Criteria:

* Under 30 years old or over 80 years old
* Is pregnant or thinks she may become pregnant.
* Open wounds on breast
* Breast implants
* Any condition that impairs the ability to give informed consent

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2014-03; Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Area under the curve for distinguishing benign vs malignant lesions | 5 years
  We will compare optical-DBT vs DBT in terms of diagnosis specificity within the diagnostic population. We will base our analysis on total hemoglobin contrast which has been shown before by our group to be significantly different between malignant and benign lesions. By setting a threshold total hemoglobin ratio and comparing with the biopsy results, we can obtain a point on the receiver operating characteristic (ROC) for the selected parameter. By sliding the threshold over all possible values, we will render the full ROC curve. The area under the curve (AUC) will be calculated to compare with that of DBT.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan A Carp, PhD, Study Director — Massachusetts General Hospital; Mansi Saksena, MBBS, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Stefan Carp, Charlestown, Massachusetts, United States